CLINICAL TRIAL: NCT05675423
Title: Imaging Characterization of the Biomechanical Coupling of Brain and Skull: An Observational Study
Brief Title: Imaging Characterization of the Biomechanical Coupling of Brain and Skull
Status: Withdrawn | Type: Observational
Why Stopped: PI has retired
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Responsible Party: Sponsor
Other Study IDs: 10000736; 000736-CC
Record Dates: First submitted 2023-01-06; First posted 2023-01-09 (Actual); Last update posted 2024-10-03 (Actual); Status verified 2024-09

CONDITIONS: Traumatic Brain Injury (Tbi); Traumatic Meningeal Enhancement (Tme)
Keywords: Traumatic Meningeal Injury; Traumatic Meningeal Enhancement; Traumatic Brain Injury; Fluid Attenuated Inversion Recovery; Natural History
MeSH Terms: conditions — Brain Injuries, Traumatic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- 25 subjects with a history of TBI but no history of TMI: 25 subjects with a history of TBI but no history of TMI.
- 25 subjects with a history of TMI: 25 subjects with a history of TMI.
- 35 healthy controls: 35 healthy controls.

SUMMARY:
Background:

Traumatic brain injury (TBI) affects over 1.7 million people in the United States each year. Many cases are mild, but people with a history of TBI may have long-term symptoms; they are also known to be more susceptible to future concussions. Researchers are working to understand how TBI affects tissues in and around the brain over the long term. This natural history study will investigate how a TBI may change the stiffness of the brain and its surrounding connective tissues.

Objective:

To see how the brain and connective tissues respond to small head movements in people with and without a prior TBI.

Eligibility:

People aged 21 to 65 years with a history of TBI. People with no history of TBI are also needed.

Design:

Participants will have 1 clinic visit that will last about 4 hours.

Participants will have a physical exam. They answer questions to make sure it is safe for them to have a magnetic resonance imaging (MRI) scan of their brain.

They will have an MRI scan in 2 parts.

During the first part, participants will lie on a table that slides into a large tube. They will hear loud knocking noises. They may wear earplugs or earmuffs. They will lie still for 15 minutes at a time. They will be in the tube for about up to 75 minutes.

The second part is called magnetic resonance elastography (MRE). Participants will lie with their head on a pillow that vibrates gently. This test will take 10 minutes.

Participants will answer questions about how they feel 1 or 2 days after the procedure.

DETAILED DESCRIPTION:
Study Description:

The study will characterize the biomechanical coupling of the brain to the skull in human volunteers with and without a history of traumatic brain injury (TBI) using magnetic resonance elastography (MRE). MRE uses the MR scanner to measure the relative motion of brain and skull while the head is vibrated at specified frequencies.

Objectives:

Our objectives are:

1. Apply MRE to characterize the skull-brain interface in 25 mild TBI patients with a history of acute TME (TME+), 25 TME-patients (mild TBI patients without TME) and 25 healthy controls.
2. To determine whether local shear strain measures within the cortex during MRE are altered in TME+ subjects. Up to 10 additional healthy controls will be recruited for technical development of imaging protocols.

Endpoints:

Study endpoints are the completion of the MRE visit for each volunteer. The MRE data will be used to characterize the S-BI using the amplitudes and temporal delays of translation and rotation across the S-BI.

ELIGIBILITY:
* INCLUSION CRITERIA:

In order to be eligible to participate in this study, an individual must meet all of the following criteria:

1. Stated willingness to comply with all study procedures and availability for the duration of the study.
2. Age 21-65.
3. Deemed medically safe for study participation by the subjects attending physician
4. Within the TBI group, subjects must have a history of mild TBI at time of initial presentation, defined as Glasgow Coma Scale score of 13-15, loss of consciousness < 30 minutes, and normal structural imaging on CT. Subjects should be less than 10 years from time of injury.
5. Within the TME group, in addition to the TBI characteristics above, subjects should additionally, have presented for TME at the time of initial presentation, evaluated by postcontrast FLAIR imaging.
6. Ability of subject to understand and the willingness to sign a written informed consent document.

EXCLUSION CRITERIA:

An individual who meets any of the following criteria will be excluded from participation in this study:

1. Within the healthy control group, any history of clinically diagnosed TBI.
2. Other known conditions outside of TBI that may affect brain anatomy.
3. Inner ear problems causing dizziness.
4. Having a height or weight not supported by the MRI scanner.
5. Contraindications to MRI (e.g. pacemaker, pregnancy, claustrophobia).
6. Unwillingness to remove cosmetic metal (e.g. piercings) for the MRI.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects 21-65 years old, healthy volunteers, subjects with history of TBI but no history of TMI and subjects with a history of TMI.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2024-09-12 (Actual); Primary Completion 2024-09-12 (Actual); Study Completion 2024-09-12 (Actual)

PRIMARY OUTCOMES:
Obtain MRE images | End of study
  MRE images will be processed to estimate global differences in the amplitudes and temporal delays of translation and rotation between brain and skull. Temporal delay reflects the lag in motion between the skull and brain, with a lower delay reflecting tighter coupling of motion.

SECONDARY OUTCOMES:
Measure skull brain coupling | End of study
  Local measures of skull-brain coupling will be measured from MRE using octahedral shear strain, with a focus at the cortical surface. Shear strains reflect the ratio of deformation to its original state, with higher strains representing higher deformation. No attachments between the brain and skull would represent a pure slip condition, resulting in negligible strain and infinitely large temporal delays.

CONTACTS AND LOCATIONS:
Overall Officials: John A Butman, M.D., Principal Investigator — National Institutes of Health Clinical Center (CC)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- [Background] Chan DD, Knutsen AK, Lu YC, Yang SH, Magrath E, Wang WT, Bayly PV, Butman JA, Pham DL. Statistical Characterization of Human Brain Deformation During Mild Angular Acceleration Measured In Vivo by Tagged Magnetic Resonance Imaging. J Biomech Eng. 2018 Oct 1;140(10):1010051-10100513. doi: 10.1115/1.4040230. PMID 30029236
- [Background] Roth TL, Nayak D, Atanasijevic T, Koretsky AP, Latour LL, McGavern DB. Transcranial amelioration of inflammation and cell death after brain injury. Nature. 2014 Jan 9;505(7482):223-8. doi: 10.1038/nature12808. Epub 2013 Dec 8. PMID 24317693
- [Background] Chiara Ricciardi M, Bokkers RP, Butman JA, Hammoud DA, Pham DL, Warach S, Latour LL. Trauma-Specific Brain Abnormalities in Suspected Mild Traumatic Brain Injury Patients Identified in the First 48 Hours after Injury: A Blinded Magnetic Resonance Imaging Comparative Study Including Suspected Acute Minor Stroke Patients. J Neurotrauma. 2017 Jan 1;34(1):23-30. doi: 10.1089/neu.2015.4338. Epub 2016 Jun 10. PMID 27215444
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_000736-CC.html